CLINICAL TRIAL: NCT00606905
Title: Intravenous Immunoglobulin (IVIG) for Treatment of Unexplained Secondary Recurrent Miscarriage: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Intravenous Immunoglobulin (IVIG) for Treatment of Unexplained Secondary Recurrent Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of British Columbia (Other); University of Tennessee (Other); Sunnybrook Health Sciences Centre (Other); Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13157A; PHS M01 RR00055
Record Dates: First submitted 2008-01-23; First posted 2008-02-05 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2010-08

CONDITIONS: Miscarriage, Recurrent; Abortion, Habitual
Keywords: Recurrent miscarriage; Recurrent spontaneous abortion; Habitual abortion; IVIG; Randomized Controlled Trial
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous | interventions — Immunoglobulins, Intravenous; gamma-Globulins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): IVIG, either Gamimune N (Talecris Biotherapeutics, Inc., Clayton, NC) or Gamunex 10% (Talecris Biotherapeutics, Inc., Clayton, NC), both as a 10% solution
  Interventions: Biological: Gamimune N or Gamunex 10%
- 2 (Placebo Comparator): normal saline
  Interventions: Other: normal saline

INTERVENTIONS:
Biological: Gamimune N or Gamunex 10% — 500 mg/kg administered in the follicular phase of the menstrual cycle. With conception, infusions every four weeks until 18-20 weeks of gestation.
  Other Names: Immune Globulin Intravenous (Human), 10%, IGIV-C, 10%
  Arms: 1
Other: normal saline — equivalent volume of normal saline
  Arms: 2

SUMMARY:
Recurrent miscarriage is a prevalent reproductive problem that affects many couples who are trying to establish a family. This clinical study will evaluate the effectiveness of intravenous immunoglobulin (IVIG) in improving the live birth rate in couples who suffer from secondary recurrent miscarriage. This study will help in providing an answer to the question of whether IVIG is helpful in secondary recurrent miscarriage.

DETAILED DESCRIPTION:
The purpose of this multi-center trial is to evaluate the efficacy of IVIG in improving the ongoing pregnancy (>20 weeks of gestation) rate in couples with unexplained secondary recurrent miscarriage, and; to characterize and compare pharmacokinetic and pharmacodynamic parameters for IVIG pre-conceptually and in the 1st and 2nd trimesters of pregnancy, so that an improved IVIG dosing strategy can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Couple has a history of unexplained secondary recurrent miscarriage.
* Most recent pregnancy occurred within one year of discontinuing contraception.

Exclusion Criteria:

* Maternal IgA deficiency
* Maternal history of immunoglobulin hypersensitivity.
* Maternal contraindication to pregnancy.
* Evidence of active hepatitis or immunocompromised state in either partner.
* Concomitant use of medication(s) for treatment of recurrent miscarriage, such as but not limited to progesterone, clomiphene citrate, acetylsalicylic acid, heparin, glucocorticoids or hCG injections.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 1999-11; Primary Completion 2009-03 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Stephenson, MD, MSc, Study Chair — University of Chicago; William Kutteh, MD, PhD, Principal Investigator — The University of Tennesee; Susan Purkiss, MD, Principal Investigator — The University of British Columbia; Cliff Librach, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Stephenson MD, Kutteh WH, Purkiss S, Librach C, Schultz P, Houlihan E, Liao C. Intravenous immunoglobulin and idiopathic secondary recurrent miscarriage: a multicentered randomized placebo-controlled trial. Hum Reprod. 2010 Sep;25(9):2203-9. doi: 10.1093/humrep/deq179. Epub 2010 Jul 15. PMID 20634190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 1999 and February 2008, a total of 82 women were recruited from seven centers: University of British Columbia, University of Chicago, University of Tennessee-Memphis, University of Toronto, Ottawa University, Yale University and McMaster University.
Pre-assignment Details: Five of the 82 withdrew consent prior to group assignment.
Groups:
- IVIG: IVIG, either Gamimune N (Talecris Biotherapeutics, Inc., Clayton, NC) or Gamunex 10% (Talecris Biotherapeutics, Inc., Clayton, NC), both as a 10% solution. 500 mg/kg adminstered in the follicular phase of the menstrual cycle. With conception, infusions every four weeks until 18-20 weeks of gestation.
Period: Overall Study
Arm/Group | IVIG | Normal Saline
Started | 38 | 39
Pregnancy | 29 | 33
Completed | 23 | 24
Not Completed | 15 | 15
Not completed — No Pregnancy | 9 | 6
Not completed — Non-Index Pregnancy | 1 | 4
Not completed — Withdrew | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG | Normal Saline | Total
Number analyzed (Participants) | 23 | 24 | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (5) | 35 (4) | 36 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Pregnancies Defined as an Ongoing Pregnancy Over 20 Weeks Gestation, Per Number of Index Pregnancies
Time Frame: 20 weeks gestation
Population: 47 women who achieved an index pregnancy, defined as the first pregnancy in the study, unless it resulted in a noneuploid miscarriage, ectopic, molar pregnancy or genetic termination, were analyzed.
Measure: Number; unit: Successful pregnancies
Arm/Group | IVIG | Normal Saline
Number analyzed (Participants) | 23 | 24
Successful pregnancies | 16 | 15
Statistical Analysis 1: Comparison: IVIG vs Normal Saline; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.41 to 4.61]

ADVERSE EVENTS:
Arm/Group | IVIG | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 9/23 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG (N=23) | Normal Saline (N=24)
myalgia, headaches, nausea, fever or chills (General disorders) | 4 (5) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
gastrointestinal symptoms (Gastrointestinal disorders) | 0 (0) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No